CLINICAL TRIAL: NCT00643474
Title: PRISMA Study (Prospective, Randomized Trial on Intensive Self-Monitoring Blood Glucose Management Added Value in Non-Insulin Treated Type 2 Diabetes Mellitus Patients)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD000577; RD0107
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2010-05

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- A (Experimental)
  Interventions: Device: Accu-Chek Aviva Meter
- B (Experimental)
  Interventions: Device: Accu-Chek Aviva Meter

INTERVENTIONS:
Device: Accu-Chek Aviva Meter — 4-point daily glucose monitoring profile 3 times per week
  Arms: A
Device: Accu-Chek Aviva Meter — Frequency and timing of SMBG not specified
  Arms: B

SUMMARY:
This randomized, parallel study compares 2 groups of type 2 non-insulin treated (NIT) diabetes patients using the Accu-Chek Aviva glucometers. One group (Intensive Group) will perform a 4-point daily glucose monitoring profile 3 times a week Monnier-based. These patients will also receive specific glycemic targets and suggestions on how to reach them following lifestyle recommendations. At the same time, investigators will use SMBG results, downloaded from glucometers, to improve patients' therapy. The second group (Control Group), will follow the SMBG standard care usually adopted in their centers. To be eligible, patients do not to have performed a previous intensive SMBG management (the execution of SMBG measurements used to modify lifestyle, diet or physical activity, in a systematic/structured manner and/or to manage therapeutic approach). The anticipated duration of the trial is 12 months, and the target sample size is 1000 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 35-75 years of age
* Non-insulin treated type 2 diabetes for 1-10 years before enrollment
* Treatment with diet and oral hypoglycemic agents, or with diet only
* HbAlc of 7.0-9.0%

Exclusion Criteria:

* Type 1 diabetes
* Insulin treatment (for >7 consecutive days)
* Previous intensive SMBG management (the execution of SMBG measurements used to modify lifestyle, diet or physical activity in a systemic/structured manner and/or to manage therapeutic approach)
* impending complications of diabetes;
* serious diseases, including cardiovascular damage or limited life expectancy;
* pregnancy

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2008-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbAlc level; percentage of subjects reaching or maintaining the risk target (represented by a combination of LBGI<=2.5 together with HBGI<=5). | Visit 5 (52 weeks after Visit 1 +/- 2 weeks).

SECONDARY OUTCOMES:
Changes in HBGI & LBGI; blood glucose test frequency, blood glucose profile, diabetes therapy, urinary 8-isoPGF2alpha, blood pressure, creatinine clearance, lipid profile & BMI; QoL & Locus of Control analysis; hypoglycemic episodes; study-related SAEs. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Marino, Study Director — Roche Diagnostics S.p.A.
Locations (39):
- Italy (39):
  - Alessandria
  - Ancona
  - Asti
  - Bari
  - Bassano del Grappa
  - Bergamo
  - Cagliari
  - Catania
  - Catanzaro
  - Fermo
  - Foggia
  - Forlì
  - Genova
  - Lanusei
  - Mariano Comense
  - Messina
  - Milan
  - Monfalcone
  - Napoli
  - Olbia
  - Padua
  - Palermo
  - Perugia
  - Pescara
  - Prato
  - Quartu S. Elena - Cagliari
  - Ravenna
  - Roma
  - Rome
  - Rovigo
  - S. Benedetto Del Tronto (AP)
  - Salerno
  - Siena
  - Terni
  - Torino
  - Treviso
  - Trieste
  - Udine
  - Vicenza

REFERENCES:
- [Derived] Russo GT, Scavini M, Acmet E, Bonizzoni E, Bosi E, Giorgino F, Tiengo A, Cucinotta D. The Burden of Structured Self-Monitoring of Blood Glucose on Diabetes-Specific Quality of Life and Locus of Control in Patients with Noninsulin-Treated Type 2 Diabetes: The PRISMA Study. Diabetes Technol Ther. 2016 Jul;18(7):421-8. doi: 10.1089/dia.2015.0358. Epub 2016 Jun 21. PMID 27327185
- [Derived] Bosi E, Scavini M, Ceriello A, Cucinotta D, Tiengo A, Marino R, Bonizzoni E, Giorgino F; PRISMA Study Group. Intensive structured self-monitoring of blood glucose and glycemic control in noninsulin-treated type 2 diabetes: the PRISMA randomized trial. Diabetes Care. 2013 Oct;36(10):2887-94. doi: 10.2337/dc13-0092. Epub 2013 Jun 4. PMID 23735724
- [Derived] Scavini M, Bosi E, Ceriello A, Giorgino F, Porta M, Tiengo A, Vespasiani G, Bottalico D, Marino R, Parkin C, Bonizzoni E, Cucinotta D. Prospective, randomized trial on intensive SMBG management added value in non-insulin-treated T2DM patients (PRISMA): a study to determine the effect of a structured SMBG intervention. Acta Diabetol. 2013 Oct;50(5):663-72. doi: 10.1007/s00592-011-0357-y. Epub 2011 Dec 22. PMID 22189755